CLINICAL TRIAL: NCT02302144
Title: A Multifactorial Exercise Program to Reduce Falls in People With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Theresa D Ellis, Assistant Professor and Director of Center for Neurorehabilitation, Boston University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BU-SAR-BAL
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Parkinson Disease
Keywords: Postural Instability (falling); Gait Disturbances (e.g., freezing); Bradykinesia (slowness of movement), rigidity
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation; Hypokinesia; Muscle Rigidity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Multi-Ex-PD (Experimental): Immediately following enrollment, subjects will participate in a group balance and strengthening program (Multi-Ex-PD) 2x/week for 90 minutes over 3 months within the Center for Neurorehabilitation at Sargent College. Each of the exercises consists of a progression which ranges from less challenging to more challenging. The program will be individualized to the subject to appropriately match their abilities. Each subject will be progressed to a more challenging exercise once specific criteria are met. Resistance for the strengthening exercises will be applied using weighted vests.
  Interventions: Behavioral: Balance & Strengthening Exercises
- Late Multi-Ex-PD (Experimental): Three months after enrollment, subjects will participate in a group balance and strengthening program (Multi-Ex-PD) 2x/week for 90 minutes over 3 months within the Center for Neurorehabilitation at Sargent College. Each of the exercises consists of a progression which ranges from less challenging to more challenging. The program will be individualized to the subject to appropriately match their abilities. Each subject will be progressed to a more challenging exercise once specific criteria are met. Resistance for the strengthening exercises will be applied using weighted vests.
  Interventions: Behavioral: Balance & Strengthening Exercises

INTERVENTIONS:
Behavioral: Balance & Strengthening Exercises — Progressive balance and strengthening exercises conducted in a group format yet tailored to each individual

SUMMARY:
The primary objective of this study is to investigate the effects of a theoretically driven, highly challenging exercise program (balance and strengthening exercises) in reducing fall rate, improving balance and reducing fear of falling in persons with Parkinson's disease.

In this pilot, randomized, cross-over study, 32 participants with Parkinson disease will be randomly assigned to either an early start (immediately following enrollment) or late start (3 months after enrollment) multifactorial exercise program which will meet 2 times per week for 1.5 hours over 3 months. The exercise program will consist of balance and strengthening exercises which will be individualized depending on the ability of each participant. Fall rate, balance, walking ability, fear of falling, mood, anxiety, and quality of life will be measured prior to the start, at 3 months and 6 months after enrollment. Subjects will be enrolled for 6-7 months.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of idiopathic Parkinson's disease (using UK Brain Bank Criteria)
* have a Hoehn & Yahr stage of 2-4 during the "ON" state
* Mini mental status score > 26
* be 40 years of age or older, so as to represent the typical age range of PD
* be on a stable dose of Parkinson's medications for at least 2 weeks prior to study onset and during the 3 month study period.
* have experienced at least one fall in the past 3 months and greater or equal to 2 falls in the past one-year (A fall was defined as an unexpected event where the person inadvertently came to rest on the ground or other lower level not due to a major intrinsic or extrinsic event)
* able to walk without physical assistance or an assistive device for at least 5 continuous minutes
* able to understand, communicate with and be understood by recruitment personnel
* able to attend the exercise program twice per week at Sargent College
* be interested in participating and provide informed consent

Exclusion Criteria:

* have a diagnosis of atypical Parkinsonism
* have a Hoehn & Yahr stage of 1 or 5
* have had previous surgical management of PD (i.e., deep brain stimulation surgery; pallidotomy)
* serious co-morbidities that may interfere with ability to participate in an exercise program (i.e., musculoskeletal, cardiovascular, and neurological (other than Parkinson's))
* be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Falls Diary | 6-7 Months
  Subjects will be asked to record each falling episode in the falls diary at the time of the fall or as soon as possible in relation to the actual time that the fall occurred. Subjects will be interviewed regarding fall episodes at each treatment session.

SECONDARY OUTCOMES:
Change in Activities-specific Balance Confidence | 6-7 Months
  Activities-specific Balance Confidence (ABC) Scale is a self-administered questionnaire in which subjects rate their level of confidence in performing a series of 16 activities.
Change in Falls Self-Efficacy | 6-7 Months
  The Falls Self-Efficacy Scale is a self-administered questionnaire in which subjects rate their level of concern about falling when performing designated activities.
Change in Balance Evaluation Systems Test (BESTest) | 6-7 Months
  The Balance Evaluation Systems Test (BESTest) is a 36 item test which is used to assess postural control / balance. Subjects are asked to perform a series of tasks such as sitting and leaning, standing on compliant and noncompliant surfaces, stepping forward, backward and to the side and walking on level and unlevel surfaces, while turning the head and while negotiating obstacles.
Change in Six-Minute Walk Test | 6-7 Months
  The six-minute walk test (6MWT) is a measure of the distance a participant walks in a 6 minute time period. The 6-minute walk test is a safe, simple and useful measure of walking ability in patients with Parkinson's disease. The test will be carried out on level, obstacle-free enclosed corridors.
Change in Freezing of Gait Questionnaire | 6-7 Months
  The Freezing of Gait Questionnaire (FOG) is a 6-item test in which the patient is interviewed and asked questions about their walking ability.
Change in Unified Parkinson's Disease Rating Scale | 6-7 Months
  Section I, II, III and IV of the Unified Parkinson's Disease Rating Scale (UPDRS) will be utilized to assess nonmotor and motor signs.
Change in Scales for Outcomes in Parkinson Disease | 6-7 Months
  The Scales for Outcomes in Parkinson Disease (SCOPA-AUT) consists of 26 items assessing autonomic function including gastrointestinal, urinary, cardiovascular, thermoregulatory, pupillomotor and sexual function.
Change in Parkinson's Disease Questionnaire-39 | 6-7 Months
  The Parkinson's Disease Questionnaire-39 (PDQ-39) is a quality of life instrument that contains 39-self-report items and was specifically developed for people with Parkinson's disease. The PDQ-39 measures the degree of healthy, competent, and satisfying participation in daily life activities.
Change in Beck Anxiety Inventory | 6-7 Months
  The Beck Anxiety Inventory (BAI) is a measure of the severity of anxiety in adolescents and adults. The items assess typical features of anxiety, and the measure.
Changes in Beck Depression Inventory Second Edition | 6-7 Months
  The Beck Depression Inventory Second Edition (BDI-II) is a measure of the severity of depression in adolescents and adults. The items target common symptoms of depression.
Changes in Penn State Worry Questionnaire | 6-7 Months
  The Penn State Worry Questionnaire (PSWQ) is a measure of the worry characteristic of generalized anxiety disorder (GAD). Specifically, this measure of pathological worry assesses three areas of worry (generality, excessiveness, and uncontrollability).
Change in Panic Disorder Severity Scale | 6-7 Months
  The Panic Disorder Severity Scale (PDSS) is a questionnaire designed to measure the overall severity of panic disorder. The items assess the severity of seven dimensions of panic disorder and associated symptoms: frequency of panic attacks, distress during panic attacks, panic-focused anticipatory anxiety, phobic avoidance of situations, phobic avoidance of physical sensations, and impairment and interference in work and social functioning.
Changes in Anxiety Sensitivity Index | 6-7 Months
  The Anxiety Sensitivity Index (ASI) is an instrument on which respondents rate the degree to which they fear negative consequences resulting from anxiety symptoms. It yields a total score, representing the global-order anxiety sensitivity factor, as well as three lower-order factor scores, representing physical, psychological, and social concerns.
Changes in Social Phobia Inventor | 6-7 Months
  The Social Phobia Inventory (SPIN) is a self-report questionnaire used to measure symptoms of social phobia (or social anxiety disorder). The SPIN specifically evaluates the spectrum of fear (e.g. fear of being embarrassed), avoidance (e.g. avoidance of parties), and physiological (e.g. blushing) symptoms associated with social phobia.
Changes in Social Interaction Anxiety Scale | 6-7 Months
  The Social Interaction Anxiety Scale (SIAS) is a self-report questionnaire used to measure general fears of social interaction and fears of being scrutinized during activities and performance tasks. The scale is intended to measure affective, behavioral, and cognitive reactions in 20 social interaction situations.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Ellis, PhD, PT, NCS, Principal Investigator — Boston University
Locations (1):
- Center for Neurorehabilitation, College of Health & Rehabilitation Sciences, Sargent College, Boston University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Gillespie LD, Robertson MC, Gillespie WJ, Lamb SE, Gates S, Cumming RG, Rowe BH. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD007146. doi: 10.1002/14651858.CD007146.pub2. PMID 19370674
- [Background] Wood BH, Bilclough JA, Bowron A, Walker RW. Incidence and prediction of falls in Parkinson's disease: a prospective multidisciplinary study. J Neurol Neurosurg Psychiatry. 2002 Jun;72(6):721-5. doi: 10.1136/jnnp.72.6.721. PMID 12023412
- [Background] Genever RW, Downes TW, Medcalf P. Fracture rates in Parkinson's disease compared with age- and gender-matched controls: a retrospective cohort study. Age Ageing. 2005 Jan;34(1):21-4. doi: 10.1093/ageing/afh203. PMID 15591480
- [Background] Melton LJ 3rd, Leibson CL, Achenbach SJ, Bower JH, Maraganore DM, Oberg AL, Rocca WA. Fracture risk after the diagnosis of Parkinson's disease: Influence of concomitant dementia. Mov Disord. 2006 Sep;21(9):1361-7. doi: 10.1002/mds.20946. PMID 16703587
- [Background] Johnell O, Melton LJ 3rd, Atkinson EJ, O'Fallon WM, Kurland LT. Fracture risk in patients with parkinsonism: a population-based study in Olmsted County, Minnesota. Age Ageing. 1992 Jan;21(1):32-8. doi: 10.1093/ageing/21.1.32. PMID 1553857
- [Background] Temlett JA, Thompson PD. Reasons for admission to hospital for Parkinson's disease. Intern Med J. 2006 Aug;36(8):524-6. doi: 10.1111/j.1445-5994.2006.01123.x. PMID 16866658
- [Background] Hely MA, Morris JG, Traficante R, Reid WG, O'Sullivan DJ, Williamson PM. The sydney multicentre study of Parkinson's disease: progression and mortality at 10 years. J Neurol Neurosurg Psychiatry. 1999 Sep;67(3):300-7. doi: 10.1136/jnnp.67.3.300. PMID 10449550
- [Background] Spottke AE, Reuter M, Machat O, Bornschein B, von Campenhausen S, Berger K, Koehne-Volland R, Rieke J, Simonow A, Brandstaedter D, Siebert U, Oertel WH, Ulm G, Dodel R. Cost of illness and its predictors for Parkinson's disease in Germany. Pharmacoeconomics. 2005;23(8):817-36. doi: 10.2165/00019053-200523080-00007. PMID 16097843
- [Background] Jacobs JV, Horak FB. Cortical control of postural responses. J Neural Transm (Vienna). 2007;114(10):1339-48. doi: 10.1007/s00702-007-0657-0. Epub 2007 Mar 29. PMID 17393068
- [Background] Bloem BR, Beckley DJ, van Dijk JG, Zwinderman AH, Remler MP, Roos RA. Influence of dopaminergic medication on automatic postural responses and balance impairment in Parkinson's disease. Mov Disord. 1996 Sep;11(5):509-21. doi: 10.1002/mds.870110506. PMID 8866492
- [Background] Chang JT, Morton SC, Rubenstein LZ, Mojica WA, Maglione M, Suttorp MJ, Roth EA, Shekelle PG. Interventions for the prevention of falls in older adults: systematic review and meta-analysis of randomised clinical trials. BMJ. 2004 Mar 20;328(7441):680. doi: 10.1136/bmj.328.7441.680. PMID 15031239
- [Background] Tinetti ME, Baker DI, McAvay G, Claus EB, Garrett P, Gottschalk M, Koch ML, Trainor K, Horwitz RI. A multifactorial intervention to reduce the risk of falling among elderly people living in the community. N Engl J Med. 1994 Sep 29;331(13):821-7. doi: 10.1056/NEJM199409293311301. PMID 8078528
- [Background] Rose DJ. Preventing falls among older adults: no "one size suits all" intervention strategy. J Rehabil Res Dev. 2008;45(8):1153-66. PMID 19235117
- [Background] Ashburn A, Fazakarley L, Ballinger C, Pickering R, McLellan LD, Fitton C. A randomised controlled trial of a home based exercise programme to reduce the risk of falling among people with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2007 Jul;78(7):678-84. doi: 10.1136/jnnp.2006.099333. Epub 2006 Nov 21. PMID 17119004
- [Background] Pickering RM, Grimbergen YA, Rigney U, Ashburn A, Mazibrada G, Wood B, Gray P, Kerr G, Bloem BR. A meta-analysis of six prospective studies of falling in Parkinson's disease. Mov Disord. 2007 Oct 15;22(13):1892-900. doi: 10.1002/mds.21598. PMID 17588236
- [Background] Ebersbach G, Edler D, Kaufhold O, Wissel J. Whole body vibration versus conventional physiotherapy to improve balance and gait in Parkinson's disease. Arch Phys Med Rehabil. 2008 Mar;89(3):399-403. doi: 10.1016/j.apmr.2007.09.031. PMID 18295614
- [Background] Horak FB. Postural orientation and equilibrium: what do we need to know about neural control of balance to prevent falls? Age Ageing. 2006 Sep;35 Suppl 2:ii7-ii11. doi: 10.1093/ageing/afl077. PMID 16926210
- [Background] Cakit BD, Saracoglu M, Genc H, Erdem HR, Inan L. The effects of incremental speed-dependent treadmill training on postural instability and fear of falling in Parkinson's disease. Clin Rehabil. 2007 Aug;21(8):698-705. doi: 10.1177/0269215507077269. PMID 17846069
- [Background] Allen NE, Canning CG, Sherrington C, Lord SR, Latt MD, Close JC, O'Rourke SD, Murray SM, Fung VS. The effects of an exercise program on fall risk factors in people with Parkinson's disease: a randomized controlled trial. Mov Disord. 2010 Jul 15;25(9):1217-25. doi: 10.1002/mds.23082. PMID 20629134
- [Background] Protas EJ, Mitchell K, Williams A, Qureshy H, Caroline K, Lai EC. Gait and step training to reduce falls in Parkinson's disease. NeuroRehabilitation. 2005;20(3):183-90. PMID 16340099
- [Background] Dorsey ER, Constantinescu R, Thompson JP, Biglan KM, Holloway RG, Kieburtz K, Marshall FJ, Ravina BM, Schifitto G, Siderowf A, Tanner CM. Projected number of people with Parkinson disease in the most populous nations, 2005 through 2030. Neurology. 2007 Jan 30;68(5):384-6. doi: 10.1212/01.wnl.0000247740.47667.03. Epub 2006 Nov 2. PMID 17082464
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Sparrow D, DeAngelis TR, Hendron K, Thomas CA, Saint-Hilaire M, Ellis T. Highly Challenging Balance Program Reduces Fall Rate in Parkinson Disease. J Neurol Phys Ther. 2016 Jan;40(1):24-30. doi: 10.1097/NPT.0000000000000111. PMID 26655100
- See also: Center for Neurorehabilitation at Boston University — http://www.bu.edu/neurorehab/research/